CLINICAL TRIAL: NCT01881191
Title: Effect of Teriflunomide (Aubagio®) on Gray Matter Pathology in Multiple Sclerosis: The 12 Months, Prospective, Observational, Single-blinded, Longitudinal Study
Brief Title: Th Effects of Aubagio on Brain Pathology in Multiple Sclerosis Studied Over 12 Months
Acronym: GZA
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Director, Buffalo Neuroimaging Analysis Center, Professor, University at Buffalo
Other Study IDs: GZ-2013-10958
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; relapsing remitting; MRI; teriflunomide; aubagio; gray matter atrophy; gray matter pathology
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum to be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Aubagio MRI: Patients with relapsing-remitting multiple sclerosis who take Aubagio will have an MRI, eye test, blood drawn, and complete a questionnaire.
  Interventions: Other: MRI
- Healthy controls: Subjects who are otherwise healthy, without neurological disorders will have an MRI, eye test, blood drawn, and complete a questionnaire.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI

SUMMARY:
This study will evaluate the effects of Aubagio on changes in the brain using MRI.

DETAILED DESCRIPTION:
Patients who take Aubagio will have an MRI, eye test, have blood taken, and complete a questionnaire on environmental risk factors to evaluate changes in the brain and on disease progression. A healthy control group will also complete the same testing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-65
* Clinically definite MS according to the Polman criteria, 52
* Relapsing MS or Healthy Control (no neurological disorders)
* Expanded Disability Status Scale (EDSS) scores ≤5.5
* Disease duration <30 years
* Normal kidney function (creatinine clearance >59 mL/min) (patients only)
* Signed informed consent
* None of the exclusion criteria

Exclusion Criteria:

* MS patients with hepatic impairment
* Nursing mothers or pregnant women who will need to undergo 12 months follow-up
* Women of childbearing potential not using reliable contraception
* Patients currently treated with leflunomide
* Serum alanine aminotransferase (ALT) >1.5 times the upper limit of normal
* A clinically significant infectious or neurological (for HC only) illness (e.g., cellulitis, abscess, pneumonia, septicemia) within 30 days prior to treatment assignment
* Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the study protocol
* Any other reasons that, in the opinion of the Investigator, indicate that the subject is unsuitable for enrollment into this study
* Other pathology related to MRI abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MS patients from the Baird MS Center, The Jacobs Neurological Institute, Department of Neurology, State University at Buffalo, NY, USA who are also taking Aubagio as their disease modifying therapy.
  Healthy controls from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The primary aim of this study is to define the effect of teriflunomide (Aubagio®) on the development of gray matter (GM) atrophy in patients with relapsing multiple sclerosis (MS) using MRI. | baseline, 6 month and 12 month

SECONDARY OUTCOMES:
The secondary objective of this study is to define the effect of teriflunomide on subcortical deep gray matter (SDGM) pathology using MRI over 12 months. | baseline, month 6 and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zivadinov, MD,PhD,FAAN, Principal Investigator — University at Buffalo
Locations (1):
- Buffalo Neuroimaging Analysis Center, Buffalo, New York, United States